CLINICAL TRIAL: NCT04003766
Title: Randomized Trial Comparing Endoscopic Ultrasound-guided Liver Biopsy vs. Percutaneous Liver Biopsy
Brief Title: Endoscopic Ultrasound vs Percutaneous Route for Liver Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AdventHealth (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 1438608
Record Dates: First submitted 2019-06-05; First posted 2019-07-01 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Liver Biopsy
Keywords: percutaneous biopsy; endoscopic guided biopsy; liver; hepatic conditions
MeSH Terms: interventions — Biopsy

STUDY DESIGN:
Intervention Model Description: This is a randomized trial comparing two methods for procuring liver biopsy: 1) EUS-guided and 2) percutaneous.
Who Masked: Care Provider
Masking Description: The pathologist will be blinded to the procedure received by the patient.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Percutaneous Biopsy (Active Comparator): The subject would undergo the standard of care procedure for a percutaneous biopsy of the liver.
  All percutaneous biopsies will be performed after administration of local anesthetic. No pre-procedure antibiotics will be administered. Subcostal or subxyphoid area will be cleaned and draped in the standard manner. 2% lidocaine solution will be injected subcutaneously using a 25-gauge needle and then administered into the subcutaneous tissue up to the liver capsule. A 16-gauge biopsy needle is inserted into the liver parenchyma under US or CT-guidance, with the location of needle placement left to the discretion of the performing radiologist. One or two core biopsy samples will be obtained. All procured specimens will be placed in a single specimen container of 10% formalin for tissue processing. When biopsy samples have been obtained, the patient will be taken to the recovery area for post-procedure monitoring.
  Interventions: Diagnostic Test: biopsy
- Endoscopic-guided Ultrasound Biopsy (Active Comparator): The subject would undergo the standard of care procedure for an endoscopic-guided biopsy of the liver.
  The left lobe of the liver is identified from the gastric lumen, EUS-guided fine needle biopsy (FNB) will be performed using a 19-gauge FNB needle, with the choice of needle type at the discretion of the performing endoscopist. Stylet will only be used to puncture the liver at the time of the first pass and then subsequently removed. No suction will be used. Fanning technique will not be used. A total of 10 to-and-fro needle movements will be performed during each pass. A total of two passes will be performed.All tissue specimens procured will be placed in a single specimen container of 10% formalin for tissue processing. When two passes are complete under EUS-guidance, the echoendoscope will be withdrawn from the patient and the patient will be taken to the recovery area for post-procedure monitoring.
  Interventions: Diagnostic Test: biopsy

INTERVENTIONS:
Diagnostic Test: biopsy — Liver biopsy (LB) is essential for the diagnosis and evaluation of a variety of hepatic conditions, such as grading/staging of chronic liver disease secondary to alcohol, non-alcoholic steatohepatitis, viral hepatitis, hemochromatosis, Wilson's disease, cholestatic liver disease, as well as in elucidating the etiology of elevation in liver tests.

SUMMARY:
This study is to evaluate and directly compare the technical success, tissue quality, diagnostic efficacy and safety profile of Percutaneous and Endoscopic Ultrasound-guided Liver Biopsy.

DETAILED DESCRIPTION:
Liver biopsy (LB) is essential for the diagnosis and evaluation of a variety of hepatic conditions, such as grading/staging of chronic liver disease secondary to alcohol, non-alcoholic steatohepatitis, viral hepatitis, hemochromatosis, Wilson's disease, cholestatic liver disease, as well as in elucidating the etiology of elevation in liver tests.1 Since it was first performed in 1883, percutaneous (PC) liver biopsy has become routine practice and is usually performed under the guidance of real-time imaging using transabdominal ultrasound (US) or computed tomography (CT).1,2 However, in recent times, liver biopsy has been increasingly performed via transgastric or transduodenal routes under endoscopic ultrasound (EUS) guidance. The perceived advantages of performing EUS-LB compared to PC-LB are the ability to simultaneously assess other organs such as common bile duct and pancreas, access to both left and right lobes of the liver and the routine use of conscious sedation during EUS procedures.3 Although single arm cohort studies and retrospective comparative studies assessing the technical success, tissue quality and safety of these different liver biopsy modalities exist, currently there are no randomized trials comparing PC and EUS-guided LB.4-7

ELIGIBILITY:
Inclusion Criteria:

1. All patients referred for liver biopsy for any reason
2. Informed consent obtained from the patient
3. ≥ 18 years old
4. Able to undergo conscious sedation for EUS procedure

Exclusion Criteria:

1. <18 years old
2. Unable to obtain informed consent from the patient
3. Medically unfit for sedation
4. Pregnant patients
5. Presence of a mass lesion in the liver requiring biopsy visualized on cross-sectional imaging
6. Irreversible coagulopathy as determined by platelet count < 50,000 mm3 or International Normalized Ratio (INR) > 1.5
7. Unable to stop anticoagulation or anti-platelet therapy for 5 days prior to the procedure
8. Hemophilia
9. Presence of an alternative etiology for elevated liver tests seen during liver biopsy, e.g. choledocholithiasis discovered during EUS examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-07-25 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2022-02-11 (Actual)

PRIMARY OUTCOMES:
Diagnostic adequacy of the tissue sample | 24 hours
  The primary outcome of the randomized trial is to compare between EUS-LB and PC-LB, the rate of procurement of diagnostically adequate specimens, defined as the presence of both maximum specimen length ≥ 25mm AND total no. of complete portal tracts ≥ 11.

SECONDARY OUTCOMES:
Specimen length | 24 hours
  Maximum specimen length in millimeters after formalin fixation will be documented.
Portal tracts | 24 hours
  The total number of complete portal tracts for each biopsy specimen will be documented.
Rates of specimen adequacy | 24 hours
  Inadequate specimen - defined as biopsy specimens from which a definitive histological diagnosis cannot be rendered by the pathologist.
Cross over | 1 week, 30 days
  The rate of crossover to the other treatment arm will be documented
Procedure duration | 24 hours
  The total length of time for the procedure will be documented in minutes.
Rate of adverse events | 24 hours, 1 week, 30 days
  The subject will be asked to report and medical records will be reviewed for any adveerse events related to the procedure.
Procedural costs | 30 days
  The subject's account will be reviewed for total costs associated with the procedure.
Pain scores | 24 hours, 1 week, 30 days
  Pain scores measured using the Visual Analog Scale (VAS) on a scale of 0 - 10 with 0 representing no pain and 10 representing the worst pain the subject has ever had; before and after biopsy has been performed.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Hasan, MD, Principal Investigator — AdventHealth
Locations (1):
- Center for Interventional Endoscopy, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD.

REFERENCES:
- [Background] Bravo AA, Sheth SG, Chopra S. Liver biopsy. N Engl J Med. 2001 Feb 15;344(7):495-500. doi: 10.1056/NEJM200102153440706. No abstract available. PMID 11172192
- [Background] Rockey DC, Caldwell SH, Goodman ZD, Nelson RC, Smith AD; American Association for the Study of Liver Diseases. Liver biopsy. Hepatology. 2009 Mar;49(3):1017-44. doi: 10.1002/hep.22742. No abstract available. PMID 19243014
- [Background] Diehl DL. Endoscopic Ultrasound-guided Liver Biopsy. Gastrointest Endosc Clin N Am. 2019 Apr;29(2):173-186. doi: 10.1016/j.giec.2018.11.002. Epub 2019 Feb 2. PMID 30846147
- [Background] Pineda JJ, Diehl DL, Miao CL, Johal AS, Khara HS, Bhanushali A, Chen EZ. EUS-guided liver biopsy provides diagnostic samples comparable with those via the percutaneous or transjugular route. Gastrointest Endosc. 2016 Feb;83(2):360-5. doi: 10.1016/j.gie.2015.08.025. Epub 2015 Aug 22. PMID 26301407
- [Background] Tublin ME, Blair R, Martin J, Malik S, Ruppert K, Demetris A. Prospective Study of the Impact of Liver Biopsy Core Size on Specimen Adequacy and Procedural Complications. AJR Am J Roentgenol. 2018 Jan;210(1):183-188. doi: 10.2214/AJR.17.17792. Epub 2017 Nov 1. PMID 29091001
- [Background] Hall TC, Deakin C, Atwal GS, Singh RK. Adequacy of percutaneous non-targeted liver biopsy under real-time ultrasound guidance when comparing the Biopince and Achieve biopsy needle. Br J Radiol. 2017 Dec;90(1080):20170397. doi: 10.1259/bjr.20170397. Epub 2017 Oct 3. PMID 28972801
- [Background] Mohan BP, Shakhatreh M, Garg R, Ponnada S, Adler DG. Efficacy and safety of EUS-guided liver biopsy: a systematic review and meta-analysis. Gastrointest Endosc. 2019 Feb;89(2):238-246.e3. doi: 10.1016/j.gie.2018.10.018. Epub 2018 Oct 31. PMID 30389469
- [Background] Wyatt J, Hubscher S, Bellamy C. Tissue pathways for liver biopsies for the investigation of medical disease and for focal lesions. London, UK: The Royal College of Pathologists; 2014.